CLINICAL TRIAL: NCT00933062
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Clinical Study to Assess the Pharmacokinetics, Safety and Tolerability of SRT2104 Administered as Single and Multiple Doses in the Fed State to Normal Healthy Male Volunteers
Brief Title: Clinical Study to Assess the Pharmacokinetics, Safety and Tolerability of SRT2104 Administered to Normal Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 113140
Record Dates: First submitted 2009-06-25; First posted 2009-07-07 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SRT2104 (Active Comparator): Subjects will receive a dose of 2.0 g SRT2104 (administered as eight 250 mg capsules) on eight occasions during the study; once as a single dose (study day 1) during Treatment Period 1, and once per day for seven consecutive days (study days 15 to 21) during Treatment Period 2.
  Interventions: Drug: SRT2104
- Placebo (Placebo Comparator): Subjects will receive placebo on eight occasions during the study; once as a single dose (study day 1) during Treatment Period 1, and once per day for seven consecutive days (study days 15 to 21) during Treatment Period 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRT2104 — 2.0 g of SRT2104 will be supplied in hard gelatin capsules each containing 250 mg SRT2104. SRT2104 will be administered within 30 minutes following the start of consumption of a standardized non-high-fat meal (approximately 650 kcal with approximately 30% of calories derived from fat). The eight capsules of SRT2104 will be orally-administered with approximately 200 mL water.
  Arms: SRT2104
Drug: Placebo — Placebo will be supplied in hard gelatine capsules containing an appropriate amount of placebo. Placebo will be administered within 30 minutes following the start of consumption of a standardized non-high-fat meal (approximately 650 kcal with approximately 30% of calories derived from fat). The eight capsules of placebo will be orally-administered with approximately 200 mL water.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the pharmacokinetic profile, safety, and tolerability of SRT2104 following administration of single and multiple oral doses (once a day for seven days) at a single dose level (2.0 g/day) to healthy male volunteers in the fed state.

DETAILED DESCRIPTION:
This is a prospective, single center, clinical study of SRT2104 administered orally; a randomized, inpatient/outpatient study to assess the safety and pharmacokinetics (PK) of SRT2104 in healthy male volunteers. Ten (10) male subjects, aged 18-60, who fulfil the inclusion/exclusion criteria, will be enrolled in this study. Subjects will receive either a dose of 2.0 g SRT2104 (administered as eight 250 mg capsules) or placebo on eight occasions during the study; once as a single dose (study day 1) during Treatment Period 1, and once per day for seven consecutive days (study days 15 to 21) during Treatment Period 2. Every administration of SRT2104 will be in the fed state (i.e. within 30 minutes following the start of consumption of a standard meal).

Subjects will be asked to sign the informed consent form at the screening visit. If eligible and willing to participate, subjects will enter into the study. Subjects will be required to attend the research unit on eight separate occasions during the study, in addition to the screening visit. Treatment Period 1 requires the subject to attend the unit for two consecutive overnight stays (Day -1 and Day 1), after which subjects will be discharged from the unit on Day 2 (following the 24 hr post-dose PK blood sample). Subjects will then be required to return to the unit for PK blood samples to be obtained on Day 3 (48 hr post-dose), Day 4 (72 hr post-dose) and Day 8 (168 hr post-dose). Following a washout period of seven days, subjects will be required to attend the unit for Treatment Period 2, which will involve eight consecutive overnight stays (Days 14 to 21), after which subjects will be discharged from the unit on Day 22 (following the 24 hr post-dose PK blood sample). Subjects will then be required to return to the unit for PK blood samples to be obtained on Day 23 (48 hr post-dose), Day 24 (72 hr post-dose) and Day 28 (168 hr post-dose).

Subjects will be randomised 8:2 (active:placebo) to receive one of the following two treatments for the duration of the study:

A. 2.0 g SRT2104 administered as eight 250 mg hard gelatin capsules B. Eight placebo capsules

Water will be restricted from 1 hour prior to dosing until 1 hour post-dose. Subjects will receive SRT2104 within 30 minutes following the start of consumption of a standardized non-high-fat meal (approximately 650 kcal with approximately 30% of calories derived from fat). A light lunch will be provided 4 hours post-dose, an evening meal approximately 8 hours post dose and a snack approximately 12 hours post dose.

Subjects will be discharged from the study on Day 28 after the 168 h PK sample has been obtained, all required safety assessments have been performed, and the subject has been confirmed clinically stable by the investigator/identified sub-investigator.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male within the age range of 18 to 60 years.
* Voluntarily sign a Research Ethics Committee (REC)-approved informed consent form to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.
* Have biochemistry, coagulation, haematology and urinalysis test results that are within normal, allowable limits (if out-of-range, must be considered clinically significant to be exclusionary) and performed within 21 days of receiving first dose of test material.
* Have a BMI (Body Mass Index) between 18.0 and 32.0 kg/m2.
* Be clear of any history of HIV and hepatitis B and C.
* Have no significant disease or clinically significant abnormal laboratory value as deemed by the investigator on the laboratory evaluations, medical history, or physical exam.
* Have a normal 12-lead ECG or an ECG with abnormality considered to be clinically insignificant.
* Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
* Agree to use an acceptable double barrier method for birth control from the Screening visit through 3 months after the last dose of test material.
* Agree to refrain from consumption of grapefruits and/or grapefruit juice from 7 days prior to Day -1 of treatment visit 1 through to the end of subject's final study visit on Day 29.

Exclusion Criteria:

* Subject has had a major illness in the past three months or any significant ongoing chronic medical illness that the Investigator would deem unfavourable for enrolment.
* Subject has renal or liver impairment.
* Subject has a history of gastro-intestinal surgery or has a current gastrointestinal disease which may influence drug absorption.
* Subject has a history, within 3 years, of drug abuse (including Benzodiazepines, opioids, amphetamine, cocaine, and THC) or a positive drug result at the Screening Visit.
* Subject smokes more than 5 cigarettes a day.
* Subject has a history of alcoholism, and/or is currently drinking more than three drinks per day [one drink is equal to one unit of alcohol (one glass of wine, half a pint of beer, one measure of a spirit)].
* Subject has participated in a clinical trial within the past three months (defined as three months from the date of last dose of an investigational medicinal product), with the exception of the SRT-2104-004 study (EudraCT number: 2008-007364-41).
* Subject has a history of difficulty in donating blood or accessibility of veins in left or right arm.
* Subject has donated blood (one unit or 350 mL) within three months prior to receiving test material.
* Subject is taking herbal products, over-the-counter medication or prescription drug therapy for which 5 times the half-life is longer than 21 days (i.e., the Screening Period) prior to enrolment into the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03-23 (Actual); Primary Completion 2009-05-12 (Actual); Study Completion 2009-05-12 (Actual)

PRIMARY OUTCOMES:
To assess the plasma pharmacokinetic profile of SRT2104 following administration of single and multiple oral doses (once a day for seven days) at a single dose level (2.0 g/day) to healthy male volunteers in the fed state. | Plasma samples will be collected pre-dose (0 h) and at the following time points following dosing on Days 1 and 21: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 48, 72 and 168 h post-dose.

SECONDARY OUTCOMES:
To assess the safety and tolerability of SRT2104 following administration of single and multiple oral doses (once a day for seven days) at a single dose level (2.0 g/day) to healthy male volunteers in the fed state. | Safety will be monitored by AEs, VS, physical exam, labs and ECGs during the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Merthyr Tydfill, Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Hoffmann E, Wald J, Lavu S, Roberts J, Beaumont C, Haddad J, Elliott P, Westphal C, Jacobson E. Pharmacokinetics and tolerability of SRT2104, a first-in-class small molecule activator of SIRT1, after single and repeated oral administration in man. Br J Clin Pharmacol. 2013 Jan;75(1):186-96. doi: 10.1111/j.1365-2125.2012.04340.x. PMID 22616762
- See also: Results for study 113140 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113140?search=study&study_ids=113140#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113140 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register